CLINICAL TRIAL: NCT03626844
Title: Maternal Outcomes Following Manual Lysis of the Placenta After Fifteen Compared to Thirty Minutes. A Randomized Controlled Trial.
Brief Title: Maternal Outcomes Following Manual Lysis of the Placenta.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources.
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0022-18EMC
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Third Stage of Delivery
Keywords: Manual Lysis, Postpartum Hemorrhage, Third Stage of Delivery.
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lysis after 15 minutes (Intervention) (Experimental): Manual Lysis of Placenta 15 minutes after Delivery.
  Interventions: Procedure: Manual Lysis of Placenta after 15 minutes (Intervention)
- Manual lysis after 30 minutes (Control) (Active Comparator): Waiting 30 minutes after delivery and then manual lysis of the placenta.
  Interventions: Procedure: Manual Lysis of Placenta after 30 minutes (Control)

INTERVENTIONS:
Procedure: Manual Lysis of Placenta after 15 minutes (Intervention) — Manual Lysis of Placenta after 15 minutes: We administer prophylactic antibiotics, under epidural analgesia, under aseptic conditions, we perform manual lysis of placenta by introducing the hand through the vagina to the uterine cavity, separating and removing the placenta.
  Other Names: Manual Lysis of Placenta after 15 minutes
  Arms: Manual Lysis after 15 minutes (Intervention)
Procedure: Manual Lysis of Placenta after 30 minutes (Control) — Manual Lysis of Placenta after 30 minutes: We administer prophylactic antibiotics, under epidural analgesia, under aseptic conditions, we perform manual lysis of placenta by introducing the hand through the vagina to the uterine cavity, separating and removing the placenta.
  Other Names: Manual Lysis of Placenta after 30 minutes
  Arms: Manual lysis after 30 minutes (Control)

SUMMARY:
Comparison of maternal outcomes following manual lysis of placenta 15 vs 30 minutes after delivery. A primary outcome of the drop in hemoglobin will be compared between the two groups. Secondary outcomes include maternal satisfaction, time to first breastfeeding, length of hospital stay, infection rate etc.

DETAILED DESCRIPTION:
Women undergoing spontaneous term vaginal delivery with epidural analgesia will be randomly assigned into one of two groups: 1. manual lysis of placenta 15 minutes after delivery. 2. waiting 30 minutes and then manual lysis of placenta. Both groups will be managed actively during the 3rd stage of delivery, including oxytocin administration and controlled cord traction. Women who develop active bleeding will be promptly treated with manual lysis and excluded from the study. Manual lysis will be performed under epidural analgesia, and prophylactic antibiotics will be administered. Primary outcome of comparison between the two groups: hemoglobin drop after delivery. Secondary outcomes include: maternal satisfaction, time to first breastfeeding, length of hospital stay, infection rate etc.

ELIGIBILITY:
Inclusion Criteria:

* Term spontaneous vaginal delivery.
* Singleton Pregnancy.
* Epidural Analgesia during delivery.
* Age between 18 and 45 years.

Exclusion Criteria:

* Active bleeding after delivery that warrants prompt removal of placenta regardless of time from delivery.
* Vacuum Extraction.
* Intrapartum Infection.
* Intrapartum fever above 38 degrees celsius.
* Wide 3rd and 4th degree perineal tears that mandate suturing under general anaesthesia.
* Thalassemia Carriers.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Drop | within 24 hours after delivery
  The difference between Hemoglobin levels before and after delivery

SECONDARY OUTCOMES:
Rate of Blood Products Given | 7 days
  Number and type of blood products given peripartum
Blood Loss | 7 days
  Calculation of estimated blood loss during delivery by accepted formulas
Febrile morbidity | within one week of delivery
  Rate of developing fever after delivery
First Nursing | 7 days
  Time until first breastfeeding
Hospital Stay | 7 days
  Length of Hospital stay in days
Maternal Satisfaction | 7 days
  Level of maternal satisfaction from the delivery process and interventions as evaluated by a numerical scale from 1 to 5 with 5 being highly satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, M.D., Study Chair — Haemek Medical Center, Afula, Israel
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deneux-Tharaux C, Macfarlane A, Winter C, Zhang WH, Alexander S, Bouvier-Colle MH; EUPHRATES Group. Policies for manual removal of placenta at vaginal delivery: variations in timing within Europe. BJOG. 2009 Jan;116(1):119-24. doi: 10.1111/j.1471-0528.2008.01996.x. PMID 19087083
- [Background] Weeks AD. The retained placenta. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):1103-17. doi: 10.1016/j.bpobgyn.2008.07.005. Epub 2008 Sep 14. PMID 18793876
- [Background] Shinar S, Schwartz A, Maslovitz S, Many A. How Long Is Safe? Setting the Cutoff for Uncomplicated Third Stage Length: A Retrospective Case-Control Study. Birth. 2016 Mar;43(1):36-41. doi: 10.1111/birt.12200. Epub 2015 Nov 10. PMID 26555024
- [Background] Tuncalp O, Souza JP, Gulmezoglu M; World Health Organization. New WHO recommendations on prevention and treatment of postpartum hemorrhage. Int J Gynaecol Obstet. 2013 Dec;123(3):254-6. doi: 10.1016/j.ijgo.2013.06.024. Epub 2013 Aug 30. PMID 24054054
- [Background] Obajimi GO, Roberts AO, Aimakhu CO, Bello FA, Olayemi O. An appraisal of retained placentae in ibadan: a five year review. Ann Ib Postgrad Med. 2009 Jun;7(1):21-5. doi: 10.4314/aipm.v7i1.64058. PMID 25161458
- [Background] Morales M, Ceysens G, Jastrow N, Viardot C, Faron G, Vial Y, Kirkpatrick C, Irion O, Boulvain M. Spontaneous delivery or manual removal of the placenta during caesarean section: a randomised controlled trial. BJOG. 2004 Sep;111(9):908-12. doi: 10.1111/j.1471-0528.2004.00228.x. PMID 15327603
- [Background] Setubal A, Clode N, Bruno-Paiva JL, Roncon I, Graca LM. Vesicouterine fistula after manual removal of placenta in a woman with previous cesarean section. Eur J Obstet Gynecol Reprod Biol. 1999 May;84(1):75-6. doi: 10.1016/s0301-2115(98)00305-4. PMID 10413231
- [Background] Akinola OI, Fabamwo AO, Oludara B, Akinola RA, Oshodi YA, Adebayo SK. Ruptured uterus and bowel injury from manual removal of placenta: a case report. Niger Postgrad Med J. 2012 Sep;19(3):181-3. PMID 23064176